CLINICAL TRIAL: NCT06206473
Title: Cognitive Dysfunctions Associated With Delirium in Critically-ill ARDS Patients: Diagnostic and Prognostic Electrophysiological Signatures
Brief Title: Cognitive Dysfunctions Associated With Delirium in Critically-ill ARDS Patients
Acronym: DeSign
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/22/0487; 2023-A00279-36 (Other: ID-RCB)
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Acute Respiratory Distress Syndrome; Delirium
Keywords: P300; N400; self-processing; semantic priming; functional connectivity
MeSH Terms: conditions — Respiratory Distress Syndrome; Delirium

STUDY DESIGN:
Intervention Model Description: single-center cohort (Intensive Care Unit of the Toulouse University Hospital), prospective, longitudinal, interventional, proof of concept study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICU patients with ARDS and delirium (Experimental): ICU patients with ARDS and delirium will be assessed twice: in the acute phase of ICU-related delirium (V1) using an mEEG battery (electrophysiological acquisition at rest and during complex cognitive stimulation), and 6 months ± 2 weeks later (V2) using a multi-domain clinical neurocognitive and psychological assessment battery.
  Interventions: Other: mEEG assessment

INTERVENTIONS:
Other: mEEG assessment — mEEG assessment (V1) will be performed at the patient's bed within 72 hours of the diagnosis of delirium. The mEEG recording, which lasts approximately 2 hours, will be performed by one of the investigators with expertise in electrophysiological acquisition. This non-invasive assessment consists of placing an EEG net on the scalp of the participants and earphones through which the auditory stimuli will be delivered.

SUMMARY:
Early cognitive assessment of critically-ill acute respiratory distress syndrome (ARDS) patients with delirium using a multidimensional electrophysiological evaluation battery (mEEG) to identify and characterize the neural correlates of cognitive dysfunctions associated with delirium (vigilance, attention, semantic and lexical processing, self-processing), and to develop a prognostic evaluation of neurocognitive and psychological disorders using an innovative non-behavioral approach.

DETAILED DESCRIPTION:
Delirium is an altered mental status associated with specific manifestations such as reduced ability to direct, focus, maintain and shift attention (DSM V criteria). The vulnerability of critically-ill ARDS patients explains the high incidence of delirium (up to 80%) in this setting. Delirium is an independent predictor of post-traumatic stress disorder, long term cognitive decline and mortality. To reduce this medical and social burden, a more complete description of delirium is needed both in terms of cognitive impairments and long term neurological and neuropsychological impact. Actually, it could be argued that the current exclusive behavioral assessment of these patients is insufficient in terms of diagnosis and prognostic assessment. In recent years, the study of consciousness has made major progress thanks to the use of innovative electrophysiological exploration methods. This work has notably allowed the development of new non-behavioral tools for the exploration of brain function in brain damaged patients in response to complex auditory stimulations (multidimensional electrophysiological battery, mEEG). In this context, the investigator team has recently demonstrated alterations in cognitive functions related to language- and self-processing in ARDS patients with severe acute respiratory syndrome (SARS)-CoV2 infection. These electrophysiological cognitive alterations were particularly marked in COVID-19 patients with delirium. Further studies are needed to disentangle the cognitive impact specifically related to delirium from that related to a severe form of COVID-19. The primary objective of this study is to identify diagnostic electrophysiological signatures of cognitive dysfunctions associated with the acute phase of delirium in critically-ill ARDS patients using a multidimensional electrophysiological assessment (mEEG) recording at rest and during auditory stimulation (first visit, V1). Secondary objectives are to characterize the impact of intensive care unit (ICU)-related delirium on neurocognitive and psychological dysfunctions observed at 6 months (second visit, V2), in order to explore the prognostic predictive value of electrophysiological data acquired during the acute phase of delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the intensive care unit with ARDS (according to Berlin criteria)
* Delirium (according to Confusion Assessment Method (CAM)-ICU criteria)
* Membership of a social security scheme
* Signed consent of the referring person
* Discontinuation of any sedative agent for ≥ 72 hours

Exclusion Criteria:

* Pre-existing psychotic disorders
* Pre-existing cognitive deficits (short Informant Questionnaire on Cognitive Decline in the Elderly (short IQCODE) ≥ 3,4)
* Recent ICU admission (> 5 days of ICU hospitalization within 6 months prior to current ICU admission)
* Patients whose delirium cannot be reliably assessed due to blindness, deafness or inability to speak French
* Patients whose life expectancy is unlikely to exceed 24 hours
* Pregnant ans breastfeeding women
* Patients under court protection
* Patients who have already participated in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Functional connectivity: weighted Symbolic Mutual Information (wSMI) measured at rest by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | Baseline
  Analysis of data from the multidimensional electrophysiological battery (mEEG) at rest during the acute phase of delirium: continuous value (between 0 and 1) of weighted Symbolic Mutual Information (wSMI)
Event-related potentials measured during auditory stimulation by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | Baseline
  Analysis of data from the multidimensional electrophysiological battery (mEEG) during auditory stimulation at the acute phase of delirium: subject's own name effect (subject's own name vs other first name) measured by spatio-temporal
Event-related potentials measured during auditory stimulation by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | Baseline
  Analysis of data from the multidimensional electrophysiological battery (mEEG) during auditory stimulation at the acute phase of delirium: local effect (local deviant tone vs local standard tone) measured by spatio-temporal clustering by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium
Event-related potentials measured during auditory stimulation by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | Baseline
  Analysis of data from the multidimensional electrophysiological battery (mEEG) during auditory stimulation at the acute phase of delirium: global effect (global deviant tone vs global standard tone) measured by spatio-temporal clustering by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium
Event-related potentials measured during auditory stimulation by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | Baseline
  • Analysis of data from the multidimensional electrophysiological battery (mEEG) during auditory stimulation at the acute phase of delirium: semantic effect (semantic unrelated words vs semantic related words) measured by spatio-temporal clustering by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium
Event-related potentials measured during auditory stimulation by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | Baseline
  • Analysis of data from the multidimensional electrophysiological battery (mEEG) at the acute phase of delirium during auditory stimulation : P3 amplitude to subject's own name stimuli (microvolts)
Event-related potentials measured during auditory stimulation by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | Baseline
  • Analysis of data from the multidimensional electrophysiological battery (mEEG) at the acute phase of delirium during auditory stimulation : P3 amplitude to local deviant tones (microvolts)
Event-related potentials measured during auditory stimulation by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | Baseline
  • Analysis of data from the multidimensional electrophysiological battery (mEEG) at the acute phase of delirium during auditory stimulation : P3 amplitude to global deviant tones (microvolts)
Event-related potentials measured during auditory stimulation by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | Baseline
  • Analysis of data from the multidimensional electrophysiological battery (mEEG) at the acute phase of delirium during auditory stimulation : N400 amplitude to semantic unrelated words (microvolts)
Event-related potentials measured during auditory stimulation by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | Baseline
  Analysis of data from the multidimensional electrophysiological battery (mEEG) at the acute phase of delirium during auditory stimulation : P3 latency to subject's own name stimuli (milliseconds)
Event-related potentials measured during auditory stimulation by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | Baseline
  Analysis of data from the multidimensional electrophysiological battery (mEEG) at the acute phase of delirium during auditory stimulation : P3 latency to local deviant tones (milliseconds)
Event-related potentials measured during auditory stimulation by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | Baseline
  • Analysis of data from the multidimensional electrophysiological battery (mEEG) at the acute phase of delirium during auditory stimulation : P3 latency to global deviant tones (milliseconds)
Event-related potentials measured during auditory stimulation by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | Baseline
  • Analysis of data from the multidimensional electrophysiological battery (mEEG) at the acute phase of delirium during auditory stimulation : N400 latency to semantic unrelated words (milliseconds)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice FERRE, MD, Principal Investigator — University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No